CLINICAL TRIAL: NCT06191263
Title: A Multicenter, Open-Label, Dose-Finding Clinical Trial to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Efficacy of RVU120 in Combination With Venetoclax in Participants With Acute Myeloid Leukemia Who Failed Prior Therapy With Ventoclax and a Hypomethylating Agent
Brief Title: Safety and Efficacy of RVU120 Combined With Venetoclax for Treatment of Relapsed/Refractory AML
Acronym: RIVER-81
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ryvu Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIVER-81
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RVU120 + Venetoclax (Experimental): RVU120 oral capsule, 125 or 250 mg administered every other day on Days 1-13 of each 21-day cycle of treatment, combined with venetoclax oral tablet, 200 or 400 mg administered once daily on Days 1-14 of each 21-day cycle of treatment
  Interventions: Drug: RVU120; Drug: Venetoclax

INTERVENTIONS:
Drug: RVU120 — RVU120 is a potent, selective inhibitor of CDK8 and its paralog CDK19
  Other Names: SEL120
Drug: Venetoclax — Venetoclax specifically binds to BCL-2, displacing proapoptotic proteins and triggering events that lead to apoptosis

SUMMARY:
The goal of this study is to assess the safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of RVU120 when administered in combination with venetoclax to adult patients with acute myeloid leukemia (AML) who are relapsed or refractory to prior therapy with venetoclax and a hypomethylating agent. The study consists of three parts. Part 1 aims to identify the doses of RVU120 and venetoclax that are considered to be safe and tolerated. Part 2 will assess the safety and efficacy of the doses selected. And Part 3 is a confirmatory cohort where patients will be treated at the same doses assessed in Part 2

DETAILED DESCRIPTION:
In Part 1 dose-escalation participants will receive escalating oral doses of RVU120 starting at 125 mg administered every other day on days 1-13, and escalating oral doses of venetoclax starting with 200 mg administered daily on days 1-14 of each 21-day cycle of treatment. The recommended doses for further study will be based on the observed safety, tolerance, PK and PD.

In Part 2, it will be assessed whether the recommended dose level from Part 1 reaches the targetted response criteria, and if reached, Part 3 will be initiated to further evaluate the efficacy and safety of the recommended doses in a larger population.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of AML (per 2022 WHO classification)
* Patients must have relapsed or refractory AML (per ELN 2022 criteria)
* Patients must have failed first-line treatment with venetoclax combined with a hypomethylating agent
* Patients must have no alternative therapeutic options likely to produce clinical benefit
* Patients must have ECOG performance status of 0 to 2
* Patients must have adequate end organ function defined as:

  1. WBC < 25 x 10(9)/L on Day 1 prior to first dose of study drug
  2. Platelet count > 10,000/mcL on Day 1 prior to first dose of study drug
  3. AST (aspartate transaminase) and ALT (alanine transaminase) ≤ 3 x ULN (upper limit of normal)
  4. Total bilirubin ≤ 3 x ULN
  5. Creatinine clearance (Cockcroft & Gault formula) ≥ 50 mL/min
  6. LVEF (left ventricular ejection fraction) ≥ 40% by electrocardiography
* Subjects must have the ability to understand and the willingness to sign a written informed consent document and complete study related procedures

Exclusion Criteria:

* APL (acute promyelocytic leukemia), the M3 subtype of AML
* Active CNS (central nervous system) leukemia
* Previous treatment with CDK8 and/or CDK19-targeted therapy
* Major surgery within 28 days prior to the first dose of study drug
* Hematopoietic stem cell transplant within 120 days prior to the first dose of study drug
* Currently pregnant or breast-feeding. Females of child bearing potential must have a negative serum pregnancy test within 72 hours prior to the first dose of study drug
* Uncontrolled intercurrent illness that could limit life expectancy or ability to complete study correlates. This includes but is not limited to:

  1. Active, Grade ≥2 acute GVHD (graft versus host disease) or requirement for systemic immunosuppressive medication for GVHD
  2. Evidence of ongoing or uncontrolled systemic bacterial, fungal or viral infection and acute inflammatory conditions (including pancreatitis)
  3. Ongoing significant liver disease such as cirrhosis, drug-induced liver injury, active hepatitis, or chronic persistent hepatitis B and/or hepatitis C
  4. Ongoing drug-induced pneumonitis
  5. Significant cardiac dysfunction, defined as myocardial infarction within 12 months prior to the first dose of study drug, NYHA (New York Heart Association) Class III or IV heart failure, uncontrolled dysrhythmias, poorly controlled angina
  6. History of ventricular arrhythmia or QTc ≥ 470 ms (Bazett's formula)
  7. Prior history of malignancies other than AML, unless disease-free for 5 years or more or prior basal cell carcinoma of the skin, non-metastatic squamous cell carcinoma of the skin, carcinoma in situ of cervix, breast or bladder, and incidental histological finding of prostate cancer (TMN stage T1a or T1b)
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RVU120 and/or venetoclax
* Taking any medications, herbal supplements, or other substances (including smoking( that are known to be strong inhibitors or moderate/strong inducers or sensitive substrates of CYP1A2
* Taking any medications, over-the-counter medications, foods or herbal supplements that are known to be strong or moderate inhibitors of CYP3A4 or P-gp (P-glycoprotein)
* Known allergy or hypersensitivity to any component of RVU120 or venetoclax formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
(Part 1) recommended doses of RVU120 and venetoclax for further study | approx. 12 months
  Incidence and severity of toxicities and number of dose limiting toxicities per dose cohort
(Parts 2 & 3) CR/CRh rate (Complete Remission/Complete Remission with incomplete Hematologic Recovery) | approx. 36 months
  Preliminary efficacy of RVU120 combined with venetoclax to recommended doses from Part 1. A response of CRh is defined as bone marrow with <5% blasts, peripheral blood neutrophil count >0.5 x 10(3)/mcL, and peripheral blood platelet count of >0.5 x 10(5)/mcL

SECONDARY OUTCOMES:
Incidence and severity of adverse events (safety and tolerability) | approx. 36 months
  Number and grade of adverse events assessed by CTCAE v5.0
Duration of response | approx. 36 months
  Time from randomization to disease progression or death in patients who achieve CR/CRh
Post baseline transfusion independence rate | approx. 36 months
  Transfusion independence is defined as a period of 56 days with no transfusion between the first dose of study drug and the last dose of study drug + 30 days. The rate of conversion of red blood cells (RBC) and platelets is defined as percentage of participants being post-baseline transfusion independent from baseline transfusion dependent
Progression-free survival | approx. 36 months
  Time from randomization until first evidence of disease progression or death
Relapse-free survival | approx. 36 months
  Number of participants alive without relapse
Overall survival | approx. 36 months
  Time from randomization to death
Percentage of patients bridged to hematopoietic stem cell transplantation | approx. 36 months
  Number of hematopoietic stem cell transplantations following response
(Parts 2 & 3) Impact of treatment on HM-PRO (hematologic malignancy specific patient reported outcome measure) | approx. 36 months
  The HM-PRO consists of two scales, Part A (Impact) that measures treatment impact on patient's health-related quality of life using a three-point Likert scale (Not at all, A little, A lot) and Part B (Signs and Symptoms) that captures the severity of disease or treatment related signs and symptoms on a three-point Likert scale (Not at all, Mild, Severe).

CONTACTS AND LOCATIONS:
Locations (37):
- France (8):
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Universitaire De Lille, Lille
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire De Nice, Nice
  - Centre Hospitalier Universitaire De Nimes, Nîmes
  - Assistance Publique Hopitaux De Paris, Paris
  - Centre Henri Becquerel, Rouen
- Italy (9):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forlì-Cesena
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Univerisity of Bologna Policlinico Sant'Orsola, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Ospedale Vito Fazzi Lecce, Lecce
  - AUSL Romagna - Ospedale S.M. Delle Croci, Ravenna
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Citta Della Salute E Della Scienza Di Torino, Turin
- Poland (10):
  - MTZ Clinical Research, Warsaw, Mazowieckie Województwo
  - Wojewodzki Szpital Specjalistyczny w Bialej Podlaskiej, Biała Podlaska
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - PRATIA Onkologia Katowice, Katowice
  - Wojewodzki Szpital Zespolony Im.L.Rydygiera w Toruniu, Torun
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Wojskowy Instytut Medyczny Panstwowy Instytut Badawczy, Warsaw
  - Specjalistyczny Szpital Im. Dra Alfreda Sokolowskiego, Wałbrzych
  - Dolnoslaskie Centrum Onkologii Pulmonologii i Hematologii, Wroclaw
  - Szpital Uniwersytecki Imienia Karola Marcinkowskiego w Zielonej Gorze Sp. z o. o., Zielona Góra
- Spain (10):
  - Hospital Del Mar, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Institut Catala D'oncologia, Barcelona
  - Hospital San Pedro De Alcantara, Cáceres
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Regional De Malaga, Málaga
  - Clinica Universidad De Navarra, Pamplona
  - University Hospital Virgen Del Rocio S.L., Seville
  - Hospital Universitario Y Politecnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No